CLINICAL TRIAL: NCT02376517
Title: Helping All Children be Safe Outdoors With Sun Protection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, June Robinson, Professor of Dermatology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: STU00200215
Record Dates: First submitted 2015-02-20; First posted 2015-03-03 (Estimated); Last update posted 2015-09-17 (Estimated); Status verified 2015-09

CONDITIONS: Children; Parents; Sun Protection
Keywords: Health Behavior; Melanin Index; Spectrophotometry; Sun Protective Clothing; Education; Primary Prevention
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Educational program (Active Comparator): Participants randomized to the intervention group will receive the educational program at the baseline visit.
  Interventions: Behavioral: Educational program
- Control (No Intervention): Participants randomized to the control group will receive the educational program at the follow-up visit.

INTERVENTIONS:
Behavioral: Educational program — The educational program consists of a short (13 pages) read-along book in English and Spanish. This book presents sun protective practices at an appropriate level for 2-6 year old children to read with their parent or caregiver. A sun protective swim shirt, which provides a sun-protection factor (SPF) of over 50, for the child will be provided. Additionally, the parent will receive weekly text message reminders to practice sun protection.
  Arms: Educational program

SUMMARY:
The purpose of this study is to test the effectiveness of a sun protection education program for children of all ethnic and racial backgrounds. Practicing sun protection in childhood can reduce the likelihood of developing skin cancer as an adult. The educational program consists of a read-along book in English and Spanish for the child to read with the parent or caregiver, text message reminders to practice sun protection, and a sun protective swim shirt for the child.

DETAILED DESCRIPTION:
Melanoma is the third most common form of cancer in adolescents and young adults in the United States. Unprotected sun exposure, particularly during childhood, is an important contributing factor in the risk of developing melanoma later in life. Targeting 2-6 year old children for primary prevention of skin cancer will minimize sun damage and may foster lifelong sun-protective behaviors that will reduce the likelihood of developing skin cancer, especially melanoma. Parental beliefs about and involvement in sun protection are important components of successful skin cancer prevention programs for children, especially young children.

This is a 12-week summer pilot study. The research seeks to develop a multicomponent sun protection program that is feasible for family practice and pediatric clinicians to introduce with anticipatory guidance during well-child visits. The program will further be implemented through a sun protection read-along book in English and Spanish and weekly text message reminders.

The sun protection program will enable behavioral change by caregivers and children of all ethnic and racial backgrounds. Testing the feasibility of delivering the intervention in a family medicine or pediatric practice will allow assessment of accrual and retention rates in a racially/ethnically diverse population, and lead the way to dissemination of good practice.

Participant in this study will be asked to complete two in-person visits at an Advocate Medical Group pediatric clinic. These visits will take place over a four to six week period. The first visit, or Baseline, may be on the same day as the child's well-visit. The second visit, or Follow-Up, will take place at the same location as the Baseline.

Participants randomized to the intervention group will receive the educational program at Baseline, whereas participants in the control group will receive the educational program during Follow-Up.

At the first visit (Baseline), the participant will:

1. Complete an anonymous short self-administered questionnaire about knowledge of sun protection and the child's sun protection habits
2. Some participants will be asked to complete a survey about cultural affiliation.
3. Receive the educational program at the first visit if randomized to the intervention group.

At the second visit (Follow-Up), the participant will:

1. Complete an anonymous short self-administered questionnaire about knowledge of sun protection and the child's sun protection habits.
2. Receive the educational program at the second visit if randomized to the control group.

At the end of each visit, the amount of melanin (pigment) in the child's skin will be measured. This involves the use of a Mexameter, a device that lightly presses on the child's arm to take a reading (picture) of how much pigment there is in his/her skin. This is neither painful nor invasive.

ELIGIBILITY:
Inclusion Criteria:

* Are at least 18 years old
* Is the parent of a 2-6 year old child attending a well-child visit
* If the parent present is female, she may be pregnant
* Are able to read in English and/or Spanish at a 6th grade level or higher
* Are able to receive text messages

Exclusion Criteria:

* Is the parent of a child less than 2 or older than 6 years old attending a visit
* Unable to read in English and/or Spanish at a 6th grade level or higher
* Unable to receive text messages
* Unable to complete study procedures with eligible child
* Unable to return to clinic for a follow-up visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2015-05; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Melanin Index at 4-6 weeks | Baseline and 4-6 Weeks
  The use of sun protection in those receiving the intervention versus the control group will be examined for correlation with melanin index of child's arm at the baseline and 4-6 week follow-up visit. Spectrophotometer measurement is the wavelength of the reflected light measured in nm. It represents the area under the curve for the all wavelengths of light, thus a reading will be expressed as (192 ±30, mean ± SD).

CONTACTS AND LOCATIONS:
Overall Officials: June K Robinson, MD, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Northwestern University Feinberg School of Medicine Department of Dermatology, Chicago, Illinois
  - Advocate Medical Group - Pediatric Clinics, Park Ridge, Illinois

REFERENCES:
- [Derived] Ho BK, Reidy K, Huerta I, Dilley K, Crawford S, Hultgren BA, Mallett KA, Turrisi R, Robinson JK. Effectiveness of a Multicomponent Sun Protection Program for Young Children: A Randomized Clinical Trial. JAMA Pediatr. 2016 Apr;170(4):334-42. doi: 10.1001/jamapediatrics.2015.4373. PMID 26857829